CLINICAL TRIAL: NCT02589483
Title: RORA (Reinforcement of Rectal Anastomosis(<10cm) With HemoPatch - Pilot Study
Brief Title: Reinforcement of Rectal Anastomosis-RORA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capio Sankt Görans Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Baxter
Record Dates: First submitted 2015-10-21; First posted 2015-10-28 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective pilot (Experimental): Patient included prospectivly will be all treated according to study protocol.The rectal anastomosis will be reinforced with HemoPatch.
  Interventions: Procedure: The rectal anastomosis will be reinforced with HemoPatch.; Device: Hemopatch

INTERVENTIONS:
Procedure: The rectal anastomosis will be reinforced with HemoPatch. — Associated with the making of the anastomosis stapled or hand sewed, the device HemoPatch will be wrapped all the way around the anastomotic circumference.
  Other Names: Hemopatch
Device: Hemopatch — The rectal anastomosis reinforced with Hemopatch

SUMMARY:
The anastomotic leaks are multivariable in its origin. The incidence varies among different centers between 4% and as high as 25%. The impact of leakage in a rectal anastomosis can be devastating for the patient and very costly for the health care system.

Prolonged hospital stay (LOS), invasive treatment and intensive care are the consequences.

The future of colorectal surgery will increasingly include older patients with increased preoperative morbidity and probably even higher risk for anastomotic leaks. which makes it suitable for reinforcing a rectal anastomosis. The goal is to shift the clinical leaks spectrum into a subclinical and therefore self-healing one.

DETAILED DESCRIPTION:
The rationale is to explore if the procedure of reinforcement with HemoPatch and bringing more mechanical strength over an extended area around the anastomosis thus lowers the incidence of clinical anastomotic leaks.

The characteristics of HemoPatch, with its structural properties such as flexibility and tissue adhesion are suitable for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Rectal surgery with anastomosis below 10 cm from anal verge

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinical anastomotic leak( elevated C reactive protein and white blood corpuscles, fever, nausea). Suspicion of a leak will be investigated with a Ct scan. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Dan Kornfeld, MD, PhD, Principal Investigator — Capio Sankt Görans Hospital
Locations (1):
- Dan Kornfeld, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bruce J, Krukowski ZH, Al-Khairy G, Russell EM, Park KG. Systematic review of the definition and measurement of anastomotic leak after gastrointestinal surgery. Br J Surg. 2001 Sep;88(9):1157-68. doi: 10.1046/j.0007-1323.2001.01829.x. PMID 11531861
- [Result] Daams F, Luyer M, Lange JF. Colorectal anastomotic leakage: aspects of prevention, detection and treatment. World J Gastroenterol. 2013 Apr 21;19(15):2293-7. doi: 10.3748/wjg.v19.i15.2293. PMID 23613621
- [Result] Dekker JW, Liefers GJ, de Mol van Otterloo JC, Putter H, Tollenaar RA. Predicting the risk of anastomotic leakage in left-sided colorectal surgery using a colon leakage score. J Surg Res. 2011 Mar;166(1):e27-34. doi: 10.1016/j.jss.2010.11.004. Epub 2010 Dec 1. PMID 21195424